CLINICAL TRIAL: NCT06455540
Title: Superior Hypogastric Plexus Block During Laparoscopic Hysterectomy
Brief Title: SUperior Hypogastric Plexus Block During Laparoscopic hysterEctomy (SUBTLE)
Acronym: SUBTLE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: E2022273
Record Dates: First submitted 2024-06-07; First posted 2024-06-12 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Hysterectomy
Keywords: Hysterectomy; Minimally invasive surgery; Quality of recovery
MeSH Terms: interventions — Nerve Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nerve block (Experimental): The superior hypogastric plexus block in this group will contain 20 mL of 0.75% ropivacaine hydrochloride.
  Interventions: Procedure: Superior hypogastric plexus block
- Placebo block (Placebo Comparator): The superior hypogastric plexus block in this group will contain 20 mL of 0.9% normal saline.
  Interventions: Procedure: Superior hypogastric plexus block

INTERVENTIONS:
Procedure: Superior hypogastric plexus block — Prior to the laparoscopic hysterectomy and any additional procedures, the superior hypogastric plexus block will be performed on all the patients. The block will contain 20 mL of 0.75% ropivacaine hydrochloride or 0.9% normal saline. The injection will be performed by tenting the presacral peritoneum, aspirating with a laparoscopic needle-tip syringe to ensure extravascular placement, and injecting the block.
  Other Names: Nerve block

SUMMARY:
This trial sest to assess the efficacy of a superior hypogastric plexus block (SHPB) for quality of recovery after a laparoscopic hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Undergoing laparoscopic hysterectomy for benign indications

Exclusion Criteria:

* Planned procedure that requires dissection of the presacral space
* Allergy to block medication (s)
* Known or suspected malignancy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2024-07-16 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery | Postoperative day 1
  The Quality of recovery (QoR) 15 is a patient-reported outcome questionnaire that measures the quality of recovery after surgery.

SECONDARY OUTCOMES:
Postoperative Pain Scores | Up to postoperative day 2
  Pain reported according to a visual rating scale from 0 to 100 points (0= no pain and 100= worst imaginable pain), which details their pain level using Visual Analog Scale (VAS) pain scores from the Brief Pain Inventory (BPI). Pain is reported on a scale of 1 to 100, and a higher score indicates greater pain intensity.
Postoperative Opioid Use | Up to postoperative day 2
  Postoperative opioid consumption during said time points
The Brief Pain Inventory (BPI) | Up to postoperative day 90
  The Brief Pain Inventory (BPI) is a self-administered questionnaire to assess the severity of pain and the impact of pain on the patient's daily functions.
The McGill Pain Questionnaire | Up to postoperative day 90
  The McGill Pain Questionnaire can be used to evaluate a person experiencing significant pain.
Incidence of Adverse events | Intraoperative (During block performance)
  Incidence of adverse events related to the plexus block (vascular puncture, hematoma, and local anesthetic systemic toxicity (LAST))
Length of stay in post-anesthesia care unit (PACU) area | Postoperative day 1
  Total time in PACU area
Quality of recovery | Up to postoperative day 2
  The Quality of recovery (QoR) 15 is a patient-reported outcome questionnaire that measures the quality of recovery after surgery.
Postoperative nausea and vomiting | Up to postoperative day 2
  number of participants with nausea or vomiting

IPD SHARING:
Plan to Share IPD: No